CLINICAL TRIAL: NCT03876197
Title: Follow-up Study of Safety and Efficacy in Subjects Who Participated in the Study of Intraglandular Mesenchymal Stem Cells in Patients With Radiation-induced Hyposalivation and Xerostomia (MESRIX)
Brief Title: Mesenchymal Stem Cells for Radiation-induced Xerostomia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Charlotte Lynggaard, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CVB2019-1; 2014-004349-29 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Radiation Toxicity; Xerostomia Due to Radiotherapy; Dry Mouth; Hyposalivation; Mesenchymal Stem Cells; Mesenchymal Stromal Cells; Long Term Adverse Effects
Keywords: Xerostomia Due to Radiotherapy
MeSH Terms: conditions — Radiation Injuries; Xerostomia; Long Term Adverse Effects

STUDY DESIGN:
Intervention Model Description: Long-term follow-up of Randomized controlled trial MESRIX
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Adipose-derived mesenchymal stem cells (Experimental): Autologous adipose-derived mesenchymal stem cells transplanted intraglandular in patients with radiation-induced hyposalivation and xerostomia
  Interventions: Biological: Autologous adipose-derived mesenchymal stem/stromal cells
- Placebo (Placebo Comparator): 2 ml placebo: Isotonic NaCl (0.9mg(ml) and human albumin (HA) 1%
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem/stromal cells — Autologous adipose-derived mesenchymal stem/stromal cells
  Arms: Autologous Adipose-derived mesenchymal stem cells
Other: Placebo — Isotonic NaCl (0,9mg/ml) and human albumin (HA) 1%
  Arms: Placebo

SUMMARY:
A prospective study for long-term follow-up (LTFU) to evaluate safety and efficacy in subjects who participated in the Phase 1/2 randomized placebo-controlled trial MESRIX.

DETAILED DESCRIPTION:
This is a LTFU study to assess the long-term and late effects of treatment with MSCs or placebo given ultrasound-guided into the submandibular glands in subjects participating in the MESRIX trial. Study participants from the MESRIX trial will be invited for a clinical visit. The visit will include medical history, an ENT examination; measurements of the saliva production by sialometry, a Magnetic resonance imaging scan (MRI) and obtaining data on the patient-reported outcome with Xerostomia Questionnaire (XQ) and Visual-Analogue-Symptomatic scale (VAS). Subjects, who are not able or willing to attend a clinical visit, will be encouraged to fill out the Questionnaires online or on paper. If a study participant has deceased, information of the cause of death will be investigated in The Danish Register of Causes of Death

ELIGIBILITY:
Inclusion Criteria:

1. Assessment of safety and treatment efficacy in subjects who were enrolled in the MESRIX Phase I/II clinical trial
2. Subjects who were treated with either autologous mesenchymal stem cells or placebo
3. Subjects who voluntarily decided to participate and signed the consent form after receiving explanations on the trial

Exclusion Criteria:

1. Subjects who were not enrolled in the MESRIX trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Serious Adverse Events (SAEs) and new chronic diseases | 5 years from randomization
  SAEs according to the ICH-GCP definition and new chronic diseases. For patients not attending the planned hospital visit consider searching The National Patient Register will be searched for registered SAEs. Number of patients
Overall survival | 5 years from randomization
  Overall survival is defined as the time from the intraglandular dose of the investigational product (MSCs or placebo) to the date of death or the date the subject is last known to be alive
Relapse of oropharyngeal cancer | 5 years from randomization
  Number of participants with relapse will be reported
New malignancies | 5 years from randomization
  Number of subjects who have new malignancies will be reported
Zoonotic Diseases | 5 years from randomization
  Number of subjects diagnosed Zoonotic Diseases will be reported

SECONDARY OUTCOMES:
Patient-reported outcome measures-Health-related quality of life (HRQoL | 5 years from randomization
  Xerostomia Questionnaire (XQ) ( Median item scores for each of the 8 questions will be reported (score range 0-10) and the XQ summary/composite score (0-100))

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lynggaard, MD, Principal Investigator — Department of Otolaryngology, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Department of Otolaryngology, University Hospital of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No